CLINICAL TRIAL: NCT04810754
Title: A Monocenter, Open Label Study to Evaluate the Safety and Efficacy of Daratumumab in Combination With Standard Background Therapy in Participants With Moderate to Severe Systemic Lupus Erythematosus
Brief Title: An Open Label Study to Evaluate Daratumumab in Participants With Moderate to Severe Systemic Lupus Erythematosus
Acronym: DARALUP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry); Labor Berlin-Charité Vivantes G.m.b.H (Unknown); German Cancer Research Center (Other); Charité Clinical Trial Office (CTO) (Unknown)
Responsible Party: Principal Investigator, Tobias Alexander, Tobias Alexander, Principal investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCM-RNT-202101; 2021-000962-14 (EudraCT Number)
Record Dates: First submitted 2021-03-11; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Daratumumab; anti-CD38; plasma cells; anti-dsDNA antibodies; lupus; CD38
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: open label, unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab subcutaneous (Experimental): open label daratumumab s.c., unblinded
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — 1800 mg per injection; 8 consecutive injections once a week; subcutaneous application in abdomen
  Other Names: DARZALEX (trade name)

SUMMARY:
This is a monocenter, open-label Phase II trial for refractory SLE patients currently on stable background immunosuppressive therapy. Treatment in this trial will be daratumumab weekly for a period of 8 weeks. This study will enroll 10 patients.

DETAILED DESCRIPTION:
This clinical trial "DARALUP" is designed to evaluate the efficacy and safety of daratumumab, a monoclonal antibody directed against CD38, in patients with systemic lupus erythematosus (SLE). This is a monocenter, open-label Phase II trial recruting SLE patients with clinical and serologic activity despite state-of-the-art immunosuppressive therapy. Treatment in this study will be Weekly daratumumab injections over a period of 8 weeks. This study will enroll 10 patients.

SLE is a sometimes severe, generalized autoimmune disease with few approved therapies to date. Therefore, the planned study offers an opportunity to identify a new, targeted therapeutic approach. Daratumumab has been studied in multiple Phase III clinical trials in patients with relapsing multiple myeloma, a plasma cell malignancy, where it demonstrated efficacy with an acceptable safety profile and has been approved since 2016 under the trade name Darzalex®. The aim is to investigate whether daratumumab provides clinically significant efficacy in SLE, another disease in which plasma cells have been shown to play a pathogenic role. Previous experience by the sponsor of this trial with the use of daratumumab in two patients with SLE suggests that one cycle of 4 weekly infusions with 16 mg/kg daratumumab was associated with a significant serologic and clinical response. In this study, a dosing regimen of 2 cycles of Darzalex is planned, with one cycle containing 4 Weekly injections. Based on the previously reported efficacy under anti-CD38 therapy, this human monoclonal antibody appears suitable for the therapy of SLE and will be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of SLE according to the 2019 EULAR/ACR Systemic Lupus Erythematosus classification criteria.
2. age between 18 and 60 years, inclusive, at consent.
3. have a body mass index (BMI) between 18 and 32 kg/m² (BMI = weight/height2), inclusive, and a body weight of no less than 35 kg.
4. demonstrate moderate to severe disease based on SLEDAI-2K score ≥ 6 observed at screening
5. SLEDAI-2K ≥ 4 for clinical features (i.e. SLEDAI excluding laboratory results) at screening
6. have a positive anti-double stranded deoxyribonucleic acid (anti-dsDNA) test, as measured by enzyme-linked immunosorbent assay (ELISA) test.
7. Failure or lack of tolerability of at least 2 previous state-of-the-art immunosuppressive drugs/immunomodulatory drugs including antimalarials (does not account for glucocorticoids).
8. if using oral corticosteroids, must be receiving this medication for at least 4 weeks and on a stable dose equivalent to an average dose of <20 mg of prednisone daily for at least 4 weeks prior to the first dose of study agent.
9. if using immunosuppressive drugs within the past 6 months, must not have exceeded the following dose levels: methotrexate 25 mg/week, azathioprine 2mg/kg/day, mycophenolate mofetil (MMF) 3g/day, or mycophenolic acid (MPA) 1440mg/day.
10. if using immunosuppressive drugs, must be using not more than 1 immunosuppressive drug (does not account for antimalarials and glucocorticoids) and not have used any additional immunosuppressive drug within the past 3 months prior to the first dose of study agent.

    Exclusion Criteria:
    * has any unstable or progressive manifestation of SLE (lupus cerebritis, optic neuritis, transverse myelitis, psychosis, uncontrolled seizures, systemic vasculitis, end-stage renal disease, rapidly progressive Class III or IV glomerulonephritis, isolated Class V lupus nephritis [i.e. without coexistent Class I, II, III, or IV nephritis], Class VI lupus nephritis, pulmonary hemorrhage, myocarditis) that is likely to warrant escalation in therapy beyond permitted background medications. Subjects requiring renal hemodialysis or peritoneal dialysis are also excluded.
    * has or has had a history of any clinically significant medical illness, or medical disorders the investigator considers significant should exclude the participant, including (but not limited to), hematological disease, immune deficiency states, respiratory disease, cardiovascular disease (including poor peripheral venous access), hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
    * has or has had a serious infection (e.g. sepsis, pneumonia, or pyelonephritis), or been hospitalized or received IV antibiotics for a serious infection during the 3 months prior to consent.
    * had major surgery, (e.g. requiring general anesthesia) within 3 months before screening.
    * has or has had an acute illness, including a common cold, within 2 weeks prior to first study treatment or has had a major illness or hospitalization within 3 months prior to consent.
    * has other inflammatory diseases that might confound the evaluations of efficacy, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis.
    * has received, is known to have received, or is suspected to have an intolerance or hypersensitivity (including delayed-type hypersensitivity) to any monoclonal antibodies or antibody fragments, is known to have allergies or clinically significant reactions to human proteins, monoclonal XML File Identifier: O1ANMGHPajQP16EY/porgcGYJv8= Page 11/23 antibodies, or antibody fragments, or to any components of the formulation used in this study, including daratumumab.
    * has received any live virus or bacterial vaccinations within 12 weeks prior to first study treatment or is expected to receive any live virus or bacterial vaccinations during the study or up to 20 weeks after last study treatment.
    * has received B cell depleting therapy within 12 months prior to first administration of the study agent (e.g. rituximab, ocrelizumab or obinutuzumab),
    * has received a therapy that inhibits B-cell activating factor (BAFF) (i.e. belimumab) within 3 months prior to first administration of the study agent.
    * has received prior experimental immunosuppressive biologic therapy for lupus (other than that described as allowed), less than 5 half-lives or 6 months, whichever is longer prior to first administration of the study agent.
    * has used oral or IV cyclophosphamide within 2 months prior to first administration of the study agent.
    * has ever been exposed to daratumumab or any anti-CD38 antibodies (e.g. TAK-079, MOR202, isatuximab).
    * has a history of, or ongoing, chronic or recurrent infection/diagnosed latent infection, including but not limited to, chronic renal infection, chronic chest infection (e.g. bronchiectasis), sinusitis, recurrent urinary tract infection (e.g. recurrent pyelonephritis), an open, draining, or infected skin wound, or an ulcer.
    * has or has had a serious infection (e.g. sepsis, pneumonia or pyelonephritis) or has been hospitalized or received IV antibiotics for a serious infection during the 3 months prior to consent.
    * Ongoing infection (requiring antibiotic treatment or fever > 38°C), including known HIV, active or chronic hepatitis B or hepatitis C.
    * has experienced a recent single dermatomal herpes zoster eruption within the past 6 months, or has a history of disseminated forms of zoster within the past 2 years prior to screening.
    * has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
    * has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening.
    * have had an opportunistic infection (e.g. pneumocystis, aspergillosis, mycobacterium avium complex).
    * has a history of malignancy within 5 years before consent (squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk of recurrence).
    * has a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location, or history of monoclonal gammopathy of undetermined significance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum anti-dsDNA antibody titers | Week 12 (i.e. 4 weeks after last daratumumab injection)
  The primary endpoint is the significant reduction of serum anti-dsDNA antibody titers after 8 repeated weekly injections of daratumumab at Week 12, i.e. 4 weeks after the last daratumumab injection, compared to baseline

SECONDARY OUTCOMES:
Assess the Incidence of Treatment-Emergent Adverse Events | through study completion, from screening up to Week 36
  Adverse Events will be as assessed and graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Clinical outcome parameter | Week 12
  Number of participants achieving Systemic Lupus Responder Index 4
SLE serology | through study completion, up to Week 36
  Evaluating the change in serum complement factor C3 levels
GC sparing | between Week 12 and Week 36
  Investigating median change of daily prednisolone dosage
Health-related quality of life | through study completion, up to Week 36
  Patient related outcome measures will be investigated, overall health assessed by Short-Form 36 Score
Health-related quality of life | through study completion, up to Week 36
  Patient related outcome measures will be investigated, Fatigue assessed by Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score

OTHER OUTCOMES:
Number and phenotype of peripheral blood leukocytes | through study completion, up to Week 36
  Assessed by flow cytometry
Change in surface expression levels of CD38 | through study completion, up to Week 36
  Assessed by flow cytometry on peripheral blood leukocyte subsets
Study drug concentration | at Week 9
  Investigate study drug maximum trough concentration (Cthrough) in plasma (only if primary endpoint is achieverd)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Alexander, MD, Principal Investigator — Charite University, Berlin, Germany

REFERENCES:
- [Background] Ostendorf L, Burns M, Durek P, Heinz GA, Heinrich F, Garantziotis P, Enghard P, Richter U, Biesen R, Schneider U, Knebel F, Burmester G, Radbruch A, Mei HE, Mashreghi MF, Hiepe F, Alexander T. Targeting CD38 with Daratumumab in Refractory Systemic Lupus Erythematosus. N Engl J Med. 2020 Sep 17;383(12):1149-1155. doi: 10.1056/NEJMoa2023325. PMID 32937047
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397